CLINICAL TRIAL: NCT06622447
Title: Beta-glucan-chitin-chitosan Polymer As a Dietary Supplement in Overweight/obese Subjects: Effects on Biomarkers of Cardiovascular Risk.
Brief Title: Beta-glucan-chitin-chitosan Polymer Supplement in Overweight/Obese Subjects: Cardiovascular Risk Biomarkers (QUITOVASC)
Acronym: QUITOVASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ICCC-14 QUITOVASC
Record Dates: First submitted 2024-09-05; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-07

CONDITIONS: Dietary Exposure
Keywords: β-Glucan; Chitin-chitosan; Fat-binding nutraceutical supplements

STUDY DESIGN:
Intervention Model Description: The intervention trial consisted of a prospective, randomized, two parallel arms, double-blinded, single-center study with 14-week of durantion, which includes 2-weeks run-in period and 12 weeks intervention period (βGluCnCs or placebo group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- βGluCnCs arm (Experimental): After a two-week run-in phase, participants (N=60) were randomly assigned to the βGluCnCs arm (N=40)
  During the intervention period, βGluCnCs arm participants received 1 stick (1.4 g/stick) of βGluCnCs product three times daily for a total of 12 weeks.
  Interventions: Dietary Supplement: βGluCnCs intervention
- Placebo arm (Experimental): After a two-week run-in phase, participants (N=60) were randomly assigned to the placebo arm (N=20)
  During the intervention period, placebo arm participants received 1 stick (1.4 g/stick) of placebo product (microcrystalline cellulose ) three times daily for a total of 12 weeks.
  Interventions: Dietary Supplement: Placebo intervention

INTERVENTIONS:
Dietary Supplement: βGluCnCs intervention — The intervention trial consisted of a prospective, randomized, two parallel arms, double-blinded, single-center study with 16-week of duration.
  Individuals were subjected to a 2 weeks run-in period. Following this, the population was randomly allocated into βGluCnCs intervention (N=40).
  During the intervention period, study participants received βGluCnCs product daily for a total of 12 weeks.
  Arms: βGluCnCs arm
Dietary Supplement: Placebo intervention — The intervention trial consisted of a prospective, randomized, two parallel arms, double-blinded, single-center study with 16-week of duration.
  Individuals were subjected to a 2 weeks run-in period. Following this, the population was randomly allocated into placebo intervention (N=20).
  During the intervention period, study participants received βGluCnCs product daily for a total of 12 weeks.
  Arms: Placebo arm

SUMMARY:
Reducing caloric intake and increasing energy expenditure as a strategy against overweight and its associated dyslipidaemia to reduce the risk of cardiovascular disease currently has a high failure rate.

For this reason, the consumption of food supplements capable of reducing intestinal fat absorption is seen as a tool of great interest.

The vast majority of existing fat-binder compounds have polymers such as chitin/chitosan as their active product. However, these are mainly derived from the exoskeleton of crustaceans, so their extraction and composition are highly variable, depending on season, geography and age.

The food supplement studied here refers to a new selective fat binder compound consisting mainly of a β-glucan/chitin/chitosan polymer (βGluQnQs), which is derived from the cell wall of the yeast Saccharomyces cerevisiae, a residue produced during brewing.

In vitro studies show that βGluCnCs has a high selective binding capacity for saturated fats with minimal impact as a ligand for omega-3 polyunsaturated fatty acids. In vivo tests in animal models and two pilot studies at clinical level corroborate the beneficial and selective effect of βGluCnCs supplementation in reducing saturated fat absorption and body weight reduction, with no adverse nutritional effects.

This study aimed to assess the impact of consuming a polysaccharide-rich compound containing β-Glucan/Chitin-Chitosan (βGluCnCs) fraction on the lipid profile and biomarkers of adipose tissue metabolism at plasma level, as well as on oxidative stress and circulating pro-inflammatory status in overweight or obese individuals, thereby reducing their cardiovascular risk.

The βGluCnCs compound was administered continuously and regularly for 12 weeks, compared to a placebo control that received microcrystalline cellulose.The effects were evaluated on lipid profile, lipoprotein subclass pattern and functionality and molecular markers associated with insulin resistance.

DETAILED DESCRIPTION:
Sample size (N=40 intervention group / N=20 placebo group) was calcultaded according results of previous studies where a sample size of less than 40 subjects in the intervention group was sufficient to show differences in the level of LDL oxidation and variables associated the degree of obesity.

The study refers to healthy adult men and women aged 25-60 years (N=60) and overweight (body mass index (BMI) 27-29.9 kg/m2) or obesity class 1 (BMI 30-34.9 kg/m2).

The study was approved by the Human Ethical Review Committee of the Hospital Sant Pau in Barcelona (register number:17/046). Informed written consent was obtained from all participants before their inclusion in the study. To confirm health status, all subjects underwent a complete physical examination conducted by the study physician.

The study lasted 14 weeks that were structured in 2 weeks of run-in and 12 weeks of intervention period divided into 4 phases of 4 weeks.

During the intervention period, study participants received 1 stick (1.4 g/stick) of βGluCnCs or placebo product (microcrystalline cellulose) three times daily for a total of 12 weeks.

Volunteers visited the centre at baseline, every 4 weeks (day 0, week 4, week 8) and at the end of the intervention period (week 12). Lifestyle and anthropometric measures were recorded, and blood samples were collected early in the morning after a 12-hour fast.

Compliance was monitored by weekly telephone contact with participants and interviews at the end of each 4-week phase of the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass index (BMI): Between 25 and 37 kg / m2

Exclusion Criteria:

* Eating disorders.
* Cardiovascular risk factors (e.g. hyperlipidemia, hypertension, and diabetes under pharmacological treatment).
* History of ischemic heart disease, arrhythmia, previous strokes, or peripheral vascular disease.
* Alcohol consumption exceeding 60 grams/day.
* Renal insufficiency (creatinine > 2mg/dl).
* Neoplasia.
* Systemic disease.
* Psychiatric illness under psychotropic drug treatment.
* Unstabilized thyroid pathology.
* Having followed or were following a hypocaloric diet or consuming dietary supplements for weight or constipation control or for cholesterol control for at least 2 months earlier to study inclusion.
* Food allergy or sensitivity.
* Pregnancy or breastfeeding.
* Currently undergoing treatment with non-steroidal anti-inflammatory drugs, antiplatelet agents, fibrates, or statins.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Adipokines Plasma Levels (Adiponectin, Leptin, Resistin) at Week 12 | Baseline and 12 weeks
  Quantification of plasma levels of adiponectin, leptin, and resistin using ELISA assays to assess changes in adipose tissue metabolism after 12 weeks of intervention.
  Unit of Measure: Concentration (ng/mL).
Chemerin (RARRES2) Plasma Levels at Week 12 | Baseline and 12 weeks
  Measurement of plasma levels of chemerin (RARRES2) using ELISA after 12 weeks of intervention to evaluate its association with adipose tissue metabolism and obesity.
  Unit of Measure: Concentration (ng/mL).
A-FABP (Adipocyte Fatty Acid-Binding Protein) Plasma Levels at Week 12 | Baseline and 12 weeks.
  Quantification of plasma levels of A-FABP using ELISA after 12 weeks of intervention, as a marker for adipose tissue metabolism.
  Unit of Measure: Concentration (ng/mL).
Fasting Blood Glucose Levels at Week 12 | Baseline and 12 weeks
  Biochemical measurement of fasting blood glucose levels after 12 weeks of intervention.
  Unit of Measure: Concentration (mg/dL).
Fasting Insulin Levels at Week 12 | Baseline and 12 weeks
  Measurement of fasting insulin levels using ELISA after 12 weeks of intervention.
  Unit of Measure: Concentration (μU/mL).
HOMA-IR (Homeostasis Model Assessment of Insulin Resistance) Index at Week 12 | Baseline and 12 weeks
  Calculation of the HOMA-IR index based on fasting insulin and fasting glucose levels after 12 weeks of intervention.
  Unit of Measure: HOMA-IR value (dimensionless)
Total Cholesterol Levels at Week 12 | Baseline and 12 weeks
  Description: Biochemical measurement of total cholesterol levels after 12 weeks of intervention.
  Unit of Measure: Concentration (mg/dL).
HDL Cholesterol Levels at Week 12 | Baseline and 12 weeks.
  Biochemical measurement of high-density lipoprotein (HDL) cholesterol levels after 12 weeks of intervention.
  Unit of Measure: Concentration (mg/dL).
LDL Cholesterol Levels at Week 12 | Baseline and 12 weeks
  Biochemical measurement of low-density lipoprotein (LDL) cholesterol levels after 12 weeks of intervention.
  Unit of Measure: Concentration (mg/dL).
Triglyceride Levels at Week 12 | Baseline and 12 weeks
  Biochemical measurement of triglyceride levels after 12 weeks of intervention. Unit of Measure: Concentration (mg/dL).

SECONDARY OUTCOMES:
Plasma Levels of Inflammatory Markers (TNF-alpha, IL-6, hsCRP) at Week 12 | Baseline and 12 weeks
  Description: Quantification of plasma levels of inflammatory markers (TNF-alpha, IL-6, and high-sensitivity C-reactive protein - hsCRP) using ELISA techniques to assess systemic inflammation.
  Unit of Measure: Concentration (pg/mL for TNF-alpha and IL-6; mg/L for hsCRP).
Plasma Lipid Peroxidation Levels (TBARS) at Week 12 | Baseline and 12 weeks
  Measurement of plasma lipid peroxidation levels using TBARS (thiobarbituric acid reactive substances) as a marker of oxidative stress.
  Unit of Measure: Concentration (μmol/L).
Plasma Antioxidant Capacity (FRAP) at Week 12 | Baseline and 12 weeks
  Measurement of plasma antioxidant capacity using the FRAP (Ferric Reducing Ability of Plasma) assay, which reflects the overall redox balance.
  Unit of Measure: Concentration (μmol/L).
Erythrocyte Superoxide Dismutase (SOD) Activity at Week 12 | Baseline and 12 weeks
  Measurement of erythrocyte superoxide dismutase (SOD) activity as a marker of enzymatic antioxidant defense.
  Unit of Measure: Activity (U/mg Hb).
LDL Resistance to Oxidation (Diene Measurement) at Week 12 | Baseline and 12 weeks
  Measurement of the resistance of low-density lipoprotein (LDL) to oxidation by assessing the formation of conjugated dienes as a marker of oxidative stress on lipoproteins.
  Unit of Measure: Concentration (μmol conjugated dienes/mg LDL).
Adverse Events (AEs) Monitoring Throughout the Study | Continuous monitoring throughout the 12-week study
  Recording and classification of adverse events (AEs), including severity grading and causal relationship to the dietary intervention. Adverse events will be documented individually for each subject and treatment group.
  Unit of Measure: Number of participants with treatment-related adverse events, severity graded according to protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Recerca-Hospital Santa Creu I Sant Pau, Barcelona, Barcelona, Spain